CLINICAL TRIAL: NCT06681571
Title: Comparison of Analgesic Effects of Subcostal Transversus Abdominis Plane Block and Rectus Sheath Block in Robotic-Assisted Laparoscopic Prostatectomies
Brief Title: Comparison of Analgesic Effects of TAP Block and RSB in RALPs
Status: Not yet recruiting | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep Koc, principal investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: ZeynepKoc002
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain
Keywords: transversus abdominis plane block; Rectus sheath block; Robot-assisted laparoscopic prostatectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAP Group: TAP block will be performed immediately after the induction of anesthesia, under ultrasond guidence.
  Interventions: Other: TAP Block
- RSB Group: RSB block will be performed immediately after the induction of anesthesia, under ultrasond guidence.
  Interventions: Other: RSB

INTERVENTIONS:
Other: TAP Block — TAP block will be performed immediately after the induction of anesthesia, under ultrasond guidence.
  Groups: TAP Group
Other: RSB — Rectus Sheath block will be performed immediately after the induction of anesthesia, under Ultrasond guidence.
  Groups: RSB Group

SUMMARY:
In this research, we aim to compare the postoperative analgesic efficacy of these two peripheral blocks in patients undergoing RALP who have received preoperative TAP block and RSB block.

DETAILED DESCRIPTION:
"Robotic-assisted laparoscopic prostatectomy (RALP) is a minimally invasive and superior technique that provides better visualization and maneuverability compared to open and laparoscopic surgical techniques. Previous studies have shown that RALP offers better postoperative oncological and physiological outcomes compared to open and laparoscopic techniques. However, RALP patients still experience pain lasting for several days postoperatively, which requires the use of analgesics such as opioids. This pain is associated with port site incisions, dissection of the prostate and surrounding tissues, bladder spasms, and transurethral catheter irritation. For this purpose, previous studies have utilized central and peripheral methods to reduce postoperative pain. Previous studies have demonstrated the analgesic benefits of TAP block and rectus sheath block in robotic-assisted radical prostatectomies. However, the number of studies in this area is limited. In this research, we aim to compare the postoperative analgesic efficacy of these two peripheral blocks in patients undergoing RALP who have received preoperative TAP block and RSB block.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-79 who underwent robotic radical prostatectomy
* Patients have ASA (American Society of Anesthesiologists) physical status score of 1-3.

Exclusion Criteria:

* Patients with an allergy to local anesthetic agents
* a platelet count below 100,000
* INR value above 2

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-79 who underwent robotic radical prostatectomy and have ASA (American Society of Anesthesiologists) physical status score of 1-3.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
post operatif analgesia consumption | postoperative 24 hous
  postoperative iv-PCA tramadole dose for the first 24 hours from iv-PCA devices.

SECONDARY OUTCOMES:
numerical rating scale (NRS) at rest | popstoperative 1. hour
  Recording the patient's pain at rest on the Numerical Rating Scale (NRS) by asking the patient
numerical rating scale (NRS) at rest | postoperative 6. hour
  Recording the patient's pain at rest on the Numerical Rating Scale (NRS) by asking the patient
numerical rating scale (NRS) at rest | postoperative 16. hour
  Recording the patient's pain at rest on the Numerical Rating Scale (NRS) by asking the patient
numerical rating scale (NRS) at rest | postoperative 24. hour
  Recording the patient's pain at rest on the Numerical Rating Scale (NRS) by asking the patient
NRS during coughing | postoperative1. hour
  The NRS for pain during coughing will be recorded by asking the patient
NRS during coughing | postoperative 6. hour
  The NRS for pain during coughing will be recorded by asking the patient
NRS during coughing | postoperative 16. hour
  The NRS for pain during coughing will be recorded by asking the patient
NRS during coughing | postoperative24. hour
  The NRS for pain during coughing will be recorded by asking the patient
postoperative nosia and vomiting (PONV) | postoperative 24 hours
  Recording the presence or absence of nausea and vomiting in the patient within the first 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Koç, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taninishi H, Matsusaki T, Morimatsu H. Transversus Abdominis Plane Block Reduced Early Postoperative Pain after Robot-assisted Prostatectomy: a Randomized Controlled Trial. Sci Rep. 2020 Feb 28;10(1):3761. doi: 10.1038/s41598-020-60687-y. PMID 32111916
- [Background] Beilstein CM, Huber M, Furrer MA, Loffel LM, Wuethrich PY, Engel D. Impact of analgesic techniques on early quality of recovery after prostatectomy: A 3-arm, randomized trial. Eur J Pain. 2022 Oct;26(9):1990-2002. doi: 10.1002/ejp.2020. Epub 2022 Aug 21. PMID 35960649
- [Background] Cosarcan SK, Gurkan Y, Manici M, Ozdemir I, Kilic M, Esen T, Ercelen O. The effect of ultrasound-guided rectus sheath block on postoperative analgesia in robot assisted prostatectomy: A randomized controlled trial. Medicine (Baltimore). 2024 Apr 26;103(17):e37975. doi: 10.1097/MD.0000000000037975. PMID 38669407